CLINICAL TRIAL: NCT03893084
Title: Women's Health Behaviors Stages of Change (Transtheoretical Model) in Preconception Period: A Randomized Control Study
Brief Title: Women's Health Behaviors Stages of Change (Transtheoretical Model) in Preconception Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Yasemin ERKAL AKSOY, Principal Investigator, Ege University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 0000-0002-7453-1205
Record Dates: First submitted 2019-03-07; First posted 2019-03-28 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Pregnancy; Women; Education
Keywords: preconception; period; education; midwfiery

STUDY DESIGN:
Intervention Model Description: The women who came to the institution were evaluated in terms of sample criteria and randomized sampling was divided into two groups. In order to be able to perform randomized sampling, random number table was obtained automatically by means of programs on internet sites by specifying the number of samples. The selection of the groups to the intervention and control group was determined by throwing a coin.
  In the data collection phase of the study, 218 women were evaluated in terms of sampling criteria. 10 women (who did not meet the criteria or refused to participate) were excluded from the study. 208 randomized women were divided into two groups as intervention and control group. During the follow-up, 15 women in the intervention group and 13 women in the control group were excluded from the study or were excluded because of pregnancy.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Preconception guidance prepared by reference to the guidelines published in the literature, women were given pre-pregnancy training.
  Interventions: Other: Pregnancy preparation training
- Control (No Intervention): The women in the control group were not given training, and routine practice was performed.

INTERVENTIONS:
Other: Pregnancy preparation training — Pregnancy preparation education; folic acid use, physical activity, nutrition, addictions counseling issues are included.
  Arms: Intervention

SUMMARY:
H0: Preconceptional preparatory training period between pregnancies with and without women is no difference in terms of changes in health behavior.

H1: Preconceptional preparatory training period between pregnancies with and without women there is a difference in terms of changes in health behavior.

DETAILED DESCRIPTION:
In order to reach for the second follow-up of women both her and her partner/mother phone number were registered.

ELIGIBILITY:
Inclusion Criteria:

* Accept to participate in the research and have signed the informed consent form,
* Being over 18 years old,
* To be literate,
* Lack of a psychological diagnosis,
* To be married,
* Having no pregnancy,
* Pregnancy is thought.

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnancy education was given to women.
Enrollment: 180 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
Women's behavior change phase | eight weeks
  The research was conducted by the researcher to evaluate the stages of behavior change related to the topics covered in preconceptional care. With the response to the questions, it is possible to determine which behavior change stage of the individuals. Women's behavioral changes were evaluated according to the five change stages on the transtheventional model. For the detailed evaluation of the individuals who are in the process of moving and maintaining, open-ended questions specific to each subject were asked.
Healthy Lifestyle Behavior Scale-II | eight weeks
  Walker et al. (1987) developed a scale to evaluate health-promoting behaviors related to the individual's healthy lifestyle. Validity and reliability study was conducted by Bahar et al. (2008). The scale consists of 52 items and all items are positive. The rating is in the form of a four-point likert (1), sometimes (2), often (3), regularly (4). The lowest score is 52 and the highest score is 208. The total score of the scale determines the healthy lifestyle behavior score. The scale consists of six sub-dimensions: Health responsibility, Physical activity, Nutrition, Spiritual development, Interpersonal relations, Stress management.
General Self-Efficacy Scale | eight weeks
  The scale was developed by Ralf Schwarzer and Mattihias Jerusalem (1995) in order to make a general assessment of perceived self-efficacy. The validity and reliability study of the scale was conducted by Aypay (2010). The scale applied to individuals aged 12 years or older consisted of 10 items. Self-sufficiency scale scores vary from 1 to 4 each. The lowest total score obtained from the scale is 10 and the highest score is 40. The high score from the self-efficacy scale indicates that the self-efficacy level is high.

CONTACTS AND LOCATIONS:
Locations (1):
- 17 Number Family Health Center, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ACOG Committee Opinion No. 442: Preconception and prenatal carrier screening for genetic diseases in individuals of Eastern European Jewish descent. Obstet Gynecol. 2009 Oct;114(4):950. doi: 10.1097/AOG.0b013e3181bd12f4. PMID 19888064
- [Background] Committee on Obstetric Practice. ACOG Committee Opinion No. 521: Update on immunization and pregnancy: tetanus, diphtheria, and pertussis vaccination. Obstet Gynecol. 2012 Mar;119(3):690-1. doi: 10.1097/AOG.0b013e31824e1327. PMID 22353979
- [Background] Atrash HK, Johnson K, Adams M, Cordero JF, Howse J. Preconception care for improving perinatal outcomes: the time to act. Matern Child Health J. 2006 Sep;10(5 Suppl):S3-11. doi: 10.1007/s10995-006-0100-4. Epub 2006 Jun 14. No abstract available. PMID 16773452
- [Background] Bhutta ZA, Das JK, Bahl R, Lawn JE, Salam RA, Paul VK, Sankar MJ, Blencowe H, Rizvi A, Chou VB, Walker N; Lancet Newborn Interventions Review Group; Lancet Every Newborn Study Group. Can available interventions end preventable deaths in mothers, newborn babies, and stillbirths, and at what cost? Lancet. 2014 Jul 26;384(9940):347-70. doi: 10.1016/S0140-6736(14)60792-3. Epub 2014 May 19. PMID 24853604
- [Background] de Weerd S, Steegers EA. The past and present practices and continuing controversies of preconception care. Community Genet. 2002;5(1):50-60. doi: 10.1159/000064631. PMID 14960900
- [Background] Walker SN, Sechrist KR, Pender NJ. The Health-Promoting Lifestyle Profile: development and psychometric characteristics. Nurs Res. 1987 Mar-Apr;36(2):76-81. PMID 3644262
- [Background] Schwarzer, R., & Jerusalem, M. (1995). Generalized Self-Efficacy scale. J. Weinman, S. Wright, & M. Johnston (Eds.), Measures in health psychology: A user's portfolio. Causal and control beliefs (pp. 35-37.).